CLINICAL TRIAL: NCT05070949
Title: Self-compassion to Reduce Diabetes Distress in Persons With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Ratanaporn Jerawatana, Principal Investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2933
Record Dates: First submitted 2021-05-15; First posted 2021-10-07 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes
Keywords: self-compassion; diabetes distress; sleep
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Self-Compassion (Experimental): Participants will meet every 2 weeks via zoom application or equivalent online meeting platforms, for 12 weeks. The sessions will be led by a clinical psychologist. The curriculum will follow mindful compassion program by Neff KD
  Interventions: Behavioral: Mindful Self-Compassion
- Wait List Control (No Intervention): Wait list control group will not participate in the MSC program during the first 12 weeks of the protocol but will be given an opportunity to participate after 12 weeks, using the same curriculum.

INTERVENTIONS:
Behavioral: Mindful Self-Compassion — Bi-weekly meeting will involve six lessons: What is Self-Compassion , Practicing Self-Compassion, Discovering your Compassionate Voice, Self-Compassion and Resilience , Self-Compassion and Burnout and Making it Count
  Arms: Mindful Self-Compassion

SUMMARY:
This study explored the effects of self-compassion intervention on diabetes distress and self-compassion.

DETAILED DESCRIPTION:
This study tests the effects of a 12-week mindful self-compassion (MSC) program in people with type 1 diabetes. Eighty participants will be randomized to the MSC program or be in a wait-list control group. Measures of primary outcome are self-compassion and diabetes- distress. Secondary outcomes are hemoglobin A1C, diabetes self-efficacy, stress and depression symptoms, and sleep quality. Outcomes will be measured at baseline, 12 weeks (end of the program) and 24 weeks (post program).

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes, age 18-30
* own computer or tablet with access to internet for meetings
* willingness to complete all 6 sessions

Exclusion criteria:

* history of self-harm or suicide attempt in the pat one year
* severe diabetic complications such as dialysis or blindness
* unstable depression, requiring ongoing medication adjustment within the last 3 months
* A1C > 11%
* Severe hypoglycemia requiring emergency room visit or hospitalization in the past 6 months
* History of Diabetic Ketoacidosis requiring hospitalization in the past 3 months
* pregnant or intend to get pregnant during the study timeframe

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Diabetes distress | baseline to 24 weeks
  Diabetes distress will be evaluated by a questionnaire. Each item is rated on a 6-point Likert scale from 1 (no problem) to 6 (serious problems).
  Scores range from 17 to 102, which the higher scores indicate the higher diabetes distress levels (A worse outcome).
Self-compassion | baseline to 24 weeks
  Self-compassion will be evaluated by a questionnaire. Each item is rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree).
  Scores range from 26 to 130, which the higher scores indicate the higher self-compassion levels (A better outcome). This outcome is reported in the mean difference of self-compassion score between two groups.

SECONDARY OUTCOMES:
Diabetes Self-efficacy | baseline to 24 weeks
  Diabetes self-efficacy will be measured by questionnaire. Each item is rated on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree).
  Scores range from 19 to 95, which the higher scores indicate the higher self-efficacy levels (A better outcome).
Hemoglobin A1C | baseline and 12 weeks
  HbA1c will be obtained by blood test.
Sleep quality | baseline to 24 weeks
  Sleep quality will be measured by a questionnaire. Each item is rated on a 4-point Likert scale from 0 (very good) to 3 (very bad).
  Scores range from 0 to 21, which the higher scores indicate poor sleep quality (A worse outcome).
Stress and depressive symptoms | baseline to 24 weeks
  stress and depressive symptoms will be measured by a questionnaire. Each item is rated on a 5-point Likert scale from 0 (never) to 4 (very often). Scores range from 0 to 40, which the higher scores indicate higher stress and depression (A worse outcome). This outcome is reported in the mean difference of stress and depression score between two groups.

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Faculty of Medicine Ramathibodi Hospital, Bangkok, Ratchatewi
  - Faculty of Medicine Chulalongkorn University, Bangkok

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fisher L, Hessler DM, Polonsky WH, Mullan J. When is diabetes distress clinically meaningful?: establishing cut points for the Diabetes Distress Scale. Diabetes Care. 2012 Feb;35(2):259-64. doi: 10.2337/dc11-1572. Epub 2012 Jan 6. PMID 22228744
- [Result] Aikens JE. Prospective associations between emotional distress and poor outcomes in type 2 diabetes. Diabetes Care. 2012 Dec;35(12):2472-8. doi: 10.2337/dc12-0181. Epub 2012 Oct 1. PMID 23033244
- [Result] Fisher L, Glasgow RE, Strycker LA. The relationship between diabetes distress and clinical depression with glycemic control among patients with type 2 diabetes. Diabetes Care. 2010 May;33(5):1034-6. doi: 10.2337/dc09-2175. Epub 2010 Feb 11. PMID 20150291
- [Result] Fisher L, Hessler D, Polonsky W, Strycker L, Masharani U, Peters A. Diabetes distress in adults with type 1 diabetes: Prevalence, incidence and change over time. J Diabetes Complications. 2016 Aug;30(6):1123-8. doi: 10.1016/j.jdiacomp.2016.03.032. Epub 2016 Apr 4. PMID 27118163
- [Result] Nicolucci A, Kovacs Burns K, Holt RI, Comaschi M, Hermanns N, Ishii H, Kokoszka A, Pouwer F, Skovlund SE, Stuckey H, Tarkun I, Vallis M, Wens J, Peyrot M; DAWN2 Study Group. Diabetes Attitudes, Wishes and Needs second study (DAWN2): cross-national benchmarking of diabetes-related psychosocial outcomes for people with diabetes. Diabet Med. 2013 Jul;30(7):767-77. doi: 10.1111/dme.12245. PMID 23711019
- [Result] Friis AM, Johnson MH, Cutfield RG, Consedine NS. Kindness Matters: A Randomized Controlled Trial of a Mindful Self-Compassion Intervention Improves Depression, Distress, and HbA1c Among Patients With Diabetes. Diabetes Care. 2016 Nov;39(11):1963-1971. doi: 10.2337/dc16-0416. Epub 2016 Jun 22. PMID 27335319
- [Result] Neff KD, Germer CK. A pilot study and randomized controlled trial of the mindful self-compassion program. J Clin Psychol. 2013 Jan;69(1):28-44. doi: 10.1002/jclp.21923. Epub 2012 Oct 15. PMID 23070875
- [Result] Tunsuchart K, Lerttrakarnnon P, Srithanaviboonchai K, Likhitsathian S, Skulphan S. Type 2 Diabetes Mellitus Related Distress in Thailand. Int J Environ Res Public Health. 2020 Mar 30;17(7):2329. doi: 10.3390/ijerph17072329. PMID 32235629
- [Result] Lotrakul M, Sumrithe S, Saipanish R. Reliability and validity of the Thai version of the PHQ-9. BMC Psychiatry. 2008 Jun 20;8:46. doi: 10.1186/1471-244X-8-46. PMID 18570645
- [Result] Sitasuwan T, Bussaratid S, Ruttanaumpawan P, Chotinaiwattarakul W. Reliability and validity of the Thai version of the Pittsburgh Sleep Quality Index. J Med Assoc Thai. 2014 Mar;97 Suppl 3:S57-67. PMID 24772581
- [Result] Wongpakaran N, Wongpakaran T. The Thai version of the PSS-10: An Investigation of its psychometric properties. Biopsychosoc Med. 2010 Jun 12;4:6. doi: 10.1186/1751-0759-4-6. PMID 20540784